CLINICAL TRIAL: NCT00814723
Title: Fluvastatin 80 mg Ret. vs Combination With Ezetimibe 10 mg in Patients With High Cardiovascular Risk
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Graz (Other)
Responsible Party: Prof. Dr. Winfried März, Medical University of Graz
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2004-002535-12
Record Dates: First submitted 2008-12-24; First posted 2008-12-25 (Estimated); Last update posted 2008-12-25 (Estimated); Status verified 2008-12

CONDITIONS: Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia | interventions — Fluvastatin; Ezetimibe

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fluvastatin (Active Comparator): Fluvastatin 80 mg MR
  Interventions: Drug: fluvastatin
- Fluvastatin + Ezetimibe (Active Comparator): Fluvastatin MR 80 mg plus Ezetimibe 10 mg
  Interventions: Drug: Fluvastatin plus ezetimibe

INTERVENTIONS:
Drug: fluvastatin — 80 mg MR, 12 weeks
  Other Names: Lescol
  Arms: Fluvastatin
Drug: Fluvastatin plus ezetimibe — fluvastatin 80 mg MR plus ezetimibe 10 mg
  Other Names: Lescol, Ezetrol
  Arms: Fluvastatin + Ezetimibe

SUMMARY:
Patients with coronary heart disease (CHD) or CHD equivalent (e. g. diabetes mellitus) often have abnormalities in lipids (hypercholesterolemia). Besides, hypercholesterolemia is an evident risk factor for atherosclerosis. Hitherto, there are only few studies of patients with primary hypercholesterolemia where the combination therapy with statins (HMG-Co-reductase inhibitors) and ezetimib was investigated. This combination therapy should be more effective in reducing low density lipoprotein cholesterol (LDL-C) and total cholesterol levels compared to monotherapy.

DETAILED DESCRIPTION:
Ezetimibe, a cholesterol-absorption inhibitor, significantly lowers low-density lipoprotein cholesterol (LDL-C) when administered in addition to statin treatment. The effect of ezetimibe on the incidence and progression of vascular disease is elusive. Therefore, our objective was to examine the effects of fluvastatin and fluvastatin plus ezetimibe on lipoprotein subfractions in patients with diabetes mellitus and/or coronary heart disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients with CHD or CHD equivalent with LDL 100-160 mg/dl
* Male or female sex
* Normal values of CK, AST and ALT
* Normal kidney function

Exclusion Criteria:

* CHD Stage III-IV
* St. p. myocardial infarction or coronary artery bypass grafting
* Pregnancy or breastfeeding
* Premenopausal women without certain contraception
* Known hypersensitivity to HMG-CoA reductase inhibitors or ezetimib

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2005-09; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Reduction in Low density lipoprotein cholesterol (LDL-C) | week 6 and 12

SECONDARY OUTCOMES:
Total cholesterol, triglycerides, HDL-C, lipoprotein subfractions, hs-CRP | week 6 and 12
adverse events, CK elevation, liver enzyme elevation | week 6, 12

CONTACTS AND LOCATIONS:
Overall Officials: Winfried März, Prof., M.D., Principal Investigator — Medical University of Graz, Synlab Medizinisches Versorgungszentrum für Labordiagnostik Heidelberg
Locations (1):
- Depart. of Internal Medicine, Medical University of Graz, Graz, Austria

REFERENCES:
- [Derived] Stojakovic T, de Campo A, Scharnagl H, Sourij H, Schmolzer I, Wascher TC, Marz W. Differential effects of fluvastatin alone or in combination with ezetimibe on lipoprotein subfractions in patients at high risk of coronary events. Eur J Clin Invest. 2010 Mar;40(3):187-94. doi: 10.1111/j.1365-2362.2009.02249.x. Epub 2010 Jan 7. PMID 20067513